CLINICAL TRIAL: NCT00915356
Title: A Double-blind, Randomised, Placebo-controlled, Multicentre, Dose-escalating Study of AZD1305 Given Intravenously for Cardioversion of Atrial Fibrillation
Brief Title: Intravenous Cardioversion of Atrial Fibrillation (AF) With AZD1305
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3191C00009; 2009-009862-15 (EudraCT No)
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation
Keywords: AZD1305; intravenous cardioversion of Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AZD1305 iv infusion
  Interventions: Drug: AZD1305
- 2 (Placebo Comparator): Placebo iv infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — Intravenous (iv) single infusion given intravenously until successful conversion of Atrial Fibrillation (AF) to Sinus Rhythm (SR) occur or for a maximum of 30 minutes
  Arms: 1
Drug: Placebo — iv single infusion given intravenously until successful conversion of Atrial Fibrillation (AF) to Sinus Rhythm (SR) occur or for a maximum of 30 minutes
  Arms: 2

SUMMARY:
This study is being carried out to see which dose of AZD1305 is safe and effective in cardioverting atrial fibrillation into normal heart rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for cardioversion of Atrial Fibrillation, ie a correction of irregular heart rhythm to normal heart rhythm
* Current episode of Atrial Fibrillation (ie irregular heart rhythm) lasting up to 3 months at randomisation
* Adequate anticoagulation according to international guidelines (ACC/AHA/ESC, 2006) or national guidelines

Exclusion Criteria:

* Potassium level below 3.8 mmol/L measured in serum or plasma
* QTcF interval >440 ms

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AZD1305 Medical Science Director, Study Director — AstraZeneca R&D, Mölndal, Sweden; Aladár Rónaszéki, Principal Investigator — Péterfy HospitalDepartment of Cardiology1076 Budapest, Péterfi Sándor str. 8-20HUNGARY
Locations (31):
- Czechia (3):
  - Research Site, Brno, CZ
  - Research Site, Prague
  - Research Site, Znojmo
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Esbjerg
  - Research Site, Svendborg
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Kecskemét
  - Research Site, Székesfehérvár
- Netherlands (4):
  - Research Site, Breda
  - Research Site, Deventer
  - Research Site, Leeuwarden
  - Research Site, Sneek
- Norway (4):
  - Research Site, Hamar
  - Research Site, Oslo
  - Research Site, Rud
  - Research Site, Tromsø
- Poland (6):
  - Research Site, Bytom
  - Research Site, Lubin
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Torun
  - Research Site, Warsaw
- Slovakia (3):
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Ružomberok
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Örebro
  - Research Site, Stockholm

REFERENCES:
- [Derived] Ronaszeki A, Alings M, Egstrup K, Gaciong Z, Hranai M, Kiraly C, Sereg M, Figatowski W, Bondarov P, Johansson S, Frison L, Edvardsson N, Berggren A. Pharmacological cardioversion of atrial fibrillation--a double-blind, randomized, placebo-controlled, multicentre, dose-escalation study of AZD1305 given intravenously. Europace. 2011 Aug;13(8):1148-56. doi: 10.1093/europace/eur120. Epub 2011 May 11. PMID 21561900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 1st patient was enrolled in the study on 25 May 2009, and the last patient completed the study on 4 December 2009. In total, 228 patients were enrolled (at 33 centres) and of the 171 patients randomised 170 patients completed the study. There was no discontinuation of the Investigational Product (IP) due to an Adverse Event (AE) in the study.
Pre-assignment Details: An enrolment visit (Visit 1) was done within 14 days before scheduled randomisation. Patients who fulfilled criteria and signed the informed consent form, could then be randomised at visit 2. The patients were to have ongoing Atrial Fibrillation with a clinical indication for cardioversion of Atrial Fibrillation (AF).
Groups:
- AZD1305 Dose Group 1: AZD1305, intravenous (IV) single infusion given intravenously until successful conversion of Atrial Fibrillation to Sinus Rhythm occur or for a maximum of 30 minutes. Infusion rate 120 ml/h, dose rate 50 mg/h.
- AZD1305 Dose Group 2: AZD1305, iv single infusion given intravenously until successful conversion of Atrial Fibrillation to Sinus Rhythm occur or for a maximum of 30 minutes. Infusion rate 120 ml/h, dose rate 101 mg/h.
- AZD1305 Dose Group 3: AZD1305, iv single infusion given intravenously until successful conversion of Atrial Fibrillation to Sinus Rhythm occur or for a maximum of 30 minutes. Infusion rate 120 ml/h, dose rate 130 mg/h.
- AZD1305 Dose Group 4: AZD1305, iv single infusion given intravenously until successful conversion of Atrial Fibrillation to Sinus Rhythm occur or for a maximum of 30 minutes. Infusion rate 120 ml/h, dose rate 180 mg/h.
- Placebo: Sodium chloride, iv single infusion given intravenously until successful conversion of Atrial Fibrillation to Sinus Rhythm occur or for a maximum of 30 minutes. Infusion rate 120 ml/h.
Period: Overall Study
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Started | 26 | 45 | 45 | 12 | 43
Completed | 25 | 45 | 45 | 12 | 43
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo | Total
Number analyzed (Participants) | 26 | 45 | 45 | 12 | 43 | 171
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 65 (9) | 65 (7) | 64 (10) | 66 (7) | 66 (9) | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 14 | 4 | 18 | 62
  Male | 17 | 28 | 31 | 8 | 25 | 109

OUTCOME MEASURES:

1. Primary Outcome: Dose-response Relationship for QTcF Interval of AZD1305
Description: QTcF-QT interval corrected for the RR interval (the time elapsing between two consecutive R waves in the electrocardiogram (ECG)) using the Fridericia formula.For each of 3 consecutive beats (5 consecutive beats if AF) a manual measurement, preferably in lead V2, of QTend intervals was done.The mean QT values of the 3 consecutive beats (5 consecutive beats if AF) were, together with RR intervals, date & time of the ECG, entered into the eCase Report Form (eCRF).The selected beats had to be marked with calipers and noted together with measured values and calculations on the print-out and signed
Time Frame: At any time post randomisation until end of Holter recording (18-24 hours post start of drug infusion).
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 25 | 45 | 45 | 12 | 42
ms | 461 [449 to 474] | 486 [476 to 495] | 490 [480 to 499] | 482 [464 to 500] | 440 [430 to 450]

2. Primary Outcome: Conversion of Atrial Fibrillation (AF) and Maintenance of Sinus Rhytm (SR)
Description: Conversion of AF to SR with maintenance of SR maintained for at least 1 minute
Time Frame: Within 90 minutes from start of infusion
Measure: Number (95% Confidence Interval); unit: Percentage of patients converted to SR
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 26 | 45 | 45 | 12 | 43
Percentage of patients converted to SR | 7.7 [0.9 to 25.1] | 17.8 [8.0 to 32.1] | 37.8 [23.8 to 53.5] | 50.0 [21.1 to 78.9] | 0.0 [0.0 to 8.2]

3. Secondary Outcome: Wide QRS Tachycardias
Description: Number of patients with wide QRS tachycardias, determined as significant arrhythmias by an Adjudication Committee (AC). The AC analysed and classified the occurrence of significant arrhythmias (other than AF or AFl) and pauses based on the 12-lead Holter reports. All pauses (≥3 sec) and all wide QRS complex tachycardias (≥3 beats, QRS ≥120 ms, and ≥120 bpm).
Time Frame: From start of study drug infusion until discharge from hospital on study day 2.
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 26 | 45 | 45 | 12 | 43
Participants | 4 [NA to NA] | 15 [NA to NA] | 16 [NA to NA] | 2 [NA to NA] | 7 [NA to NA]

4. Secondary Outcome: Heart Rhythm. Number of Participants With Early Relapse Into AF.
Description: Early relapse into AF within 5 minutes from obtaining the defined criterion for conversion to SR (i.e.1 minute in SR). Patients never converted are not included in the analysis.
Time Frame: Within 5 minutes following investigational product (IP) induced conversion, or direct current (DC) cardioversion, of AF to SR
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 24 | 34 | 40 | 9 | 34
Participants | 1 [NA to NA] | 1 [NA to NA] | 2 [NA to NA] | 0 [NA to NA] | 1 [NA to NA]

5. Secondary Outcome: Heart Rhythm. Number of Patients Remaining in SR up to 24 h Following Start of Study Drug Infusion
Time Frame: During 24 hours following start of study drug infusion
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 26 | 45 | 45 | 12 | 43
Participants | 23 [NA to NA] | 34 [NA to NA] | 36 [NA to NA] | 10 [NA to NA] | 33 [NA to NA]

6. Secondary Outcome: Heart Rhythm. Number of Patients Remaining in SR up to 13 to 18 Days Following Study Drug Infusion.
Description: Number of patients in SR at day 13-18
Time Frame: During 13 to 18 days following study drug infusion
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 25 | 45 | 45 | 12 | 43
Participants | 14 [NA to NA] | 23 [NA to NA] | 25 [NA to NA] | 7 [NA to NA] | 22 [NA to NA]

7. Secondary Outcome: Study the Relationship Between Systemic Exposure and Response, With Special Regards to Conversion of AF to SR and the Effect on the QTcF Interval.
Time Frame: Since this study is no longer intended to be part of any marketing authorisation application, the analyses addressing this objective were not conducted.
Reporting Status: Not Posted

8. Secondary Outcome: Maximal Observed Plasma Concentration of AZD1305
Description: Plasma concentration of AZD1305
Time Frame: Up to 24 hours following start of study drug infusion
Measure: Median (Full Range); unit: mol/L
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 24 | 41 | 43 | 11 | 0
mol/L | 0.521 [0.157 to 0.991] | 1.28 [0.374 to 2.97] | 1.39 [0.017 to 3.17] | 1.69 [0.873 to 3.61] |

9. Secondary Outcome: Conversion From AF to SR Within 90 Minutes From Start of Infusion in the Subgroup of Patients With Duration of Current AF Episode 10 Hours to 7 Days
Time Frame: Conversion from AF to SR within 90 minutes from start of infusion
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 3 | 5 | 7 | 1 | 5
Participants | 0 [NA to NA] | 2 [NA to NA] | 5 [NA to NA] | 1 [NA to NA] | 0 [NA to NA]

10. Secondary Outcome: Conversion From AF to SR Within 90 Minutes From Start of Infusion in the Subgroup of Patients With Duration of Current AF Episode 8 Days - 30 Days.
Description: Subgroup analysis for patients with duration of current AF episode 8 days - 30 days. Number of patients converting from AF to SR.
Time Frame: Conversion from AF to SR within 90 minutes from start of infusion
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 5 | 13 | 16 | 4 | 8
Participants | 0 [NA to NA] | 4 [NA to NA] | 6 [NA to NA] | 2 [NA to NA] | 0 [NA to NA]

11. Secondary Outcome: Conversion From AF to SR Within 90 Minutes From Start of Infusion in the Subgroup of Patients With Duration of Current AF Episode 31 Days - 3 Months
Description: Subgroup analysis for patients with duration of current AF episode 31 days - 3 months. Number of patients converting from AF to SR.
Time Frame: Conversion from AF to SR within 90 minutes from start of infusion
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 18 | 27 | 22 | 7 | 30
Participants | 2 [NA to NA] | 2 [NA to NA] | 6 [NA to NA] | 3 [NA to NA] | 0 [NA to NA]

12. Secondary Outcome: Percentage of Patients, Discharged Within 6 h (QTcF ≤500 ms) After Start of Infusion
Description: Percentage, with 95% confidence interval, of patients with QTcF≤500 ms six hours following start of study drug infusion
Time Frame: Six hours following start of study drug infusion
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 23 | 44 | 45 | 12 | 40
Percent of participants | 100.0 [85.2 to 100.0] | 95.5 [84.5 to 99.4] | 91.1 [78.8 to 97.5] | 100.0 [73.5 to 100.0] | 100.0 [91.2 to 100.0]

ADVERSE EVENTS:
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 3 | 3 | 1 | 2
Other Adverse Events (participants affected / at risk) | 5/26 | 9/45 | 8/45 | 3/12 | 5/43
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Atrial fibrillation (Cardiac disorders) | 1/26 | 1/45 | 0/45 | 0/12 | 0/43
Sinus bradycardia (Cardiac disorders) | 1/26 | 0/45 | 0/45 | 0/12 | 0/43
Cerebrovascular accident (Nervous system disorders) | 0/26 | 1/45 | 0/45 | 0/12 | 0/43
Multiple drug overdose (Injury, poisoning and procedural complications) | 0/26 | 1/45 | 0/45 | 0/12 | 0/43
Torsade de pointes (Cardiac disorders) | 0/26 | 0/45 | 1/45 | 0/12 | 0/43
Transient ischaemic attack (Nervous system disorders) | 0/26 | 0/45 | 1/45 | 0/12 | 0/43
Cardiac asthma (Cardiac disorders) | 0/26 | 0/45 | 1/45 | 0/12 | 0/43
Urinary tract infection (Infections and infestations) | 0/26 | 0/45 | 1/45 | 0/12 | 0/43
Ventricular tachycardia (Cardiac disorders) | 0/26 | 0/45 | 0/45 | 1/12 | 0/43
Presyncope (Nervous system disorders) | 0/26 | 0/45 | 0/45 | 1/12 | 0/43
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/26 | 0/45 | 0/45 | 0/12 | 1/43
Abdominal wall haematoma (Gastrointestinal disorders) | 0/26 | 0/45 | 0/45 | 0/12 | 1/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1305 Dose Group 1 (N=26) | AZD1305 Dose Group 2 (N=45) | AZD1305 Dose Group 3 (N=45) | AZD1305 Dose Group 4 (N=12) | Placebo (N=43)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 6 | 5 | 0 | 4
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Gastritis fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 2 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days